CLINICAL TRIAL: NCT03605745
Title: Minimally Invasive Prostatic Vapor Ablation - Multicenter, Single Arm Study for the Treatment of BPH in Large Prostates (Rezūm XL)
Brief Title: Minimally Invasive Prostatic Vapor Ablation for the Treatment of BPH in Large Prostates (Rezūm XL)
Acronym: Rezūm XL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decided to terminate the study due to business reasons
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3034-001
Record Dates: First submitted 2018-07-23; First posted 2018-07-30 (Actual); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: BPH With Urinary Obstruction; BPH; BPH With Urinary Obstruction With Other Lower Urinary Tract Symptoms
Keywords: BPH; Minimally Invasive; Water Vapor Therapy; Rezum

STUDY DESIGN:
Intervention Model Description: This study is a prospective, non-randomized clinical trial of subjects with benign prostatic hypertrophy (BPH).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Experimental): Prostatic Vapor Ablation with Rezum
  Interventions: Device: Prostatic Vapor Ablation

INTERVENTIONS:
Device: Prostatic Vapor Ablation — Rezūm uses the stored thermal energy in water vapor (steam) to treat the extra prostate tissue that is causing symptoms such as frequency, urgency, irregular flow, weak stream, straining and getting up at night to urinate.
  Inside a hand-held device, radiofrequency energy is applied to a few drops of water to create vapor (steam). The water vapor is injected into the prostate tissue that is blocking the flow of urine from the bladder, where it immediately turns back to water, releasing the energy stored in the vapor into the cell membranes. At this point, the cells are gently and immediately damaged, causing cell death. Over time, the body absorbs the treated tissue through its natural healing response.
  Other Names: Rezum; Water Vapor Ablation

SUMMARY:
Prospective, multicenter, single arm clinical trial designed to evaluate the safety of the Rezūm System in treating subjects with symptomatic BPH for prostate sizes >80cm3 and ≤150 cm3.

DETAILED DESCRIPTION:
A prospective, multicenter, single arm clinical trial designed to evaluate the safety of the Rezūm System in treating subjects with symptomatic BPH for prostate sizes >80cm3 and ≤150 cm3.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects ≥ 50 years of age who have symptomatic BPH.
2. International Prostate Symptom Score (IPSS) score ≥ 13.
3. Peak urinary flow rate (Qmax): ≥ 5ml/sec to ≤ 12 ml/sec with minimum voided volume of ≥ 125 ml.
4. Post-void residual (PVR) ≤300 ml.
5. Prostate volume >80 cm3 to ≤150 cm3

Exclusion Criteria:

Urology:

1. Any prior invasive prostate intervention (e.g., "Radiofrequency" thermotherapy, balloon, microwave thermotherapy, "Prostatic Urethral Lift", "Transurethral Resection", or laser) or other surgical interventions of the prostate.
2. Undergone a prostate biopsy within 60 days prior to the scheduled treatment date or has an imminent need for surgery.
3. Verified acute bacterial prostatitis within last 12 months documented by culture.
4. Active or history of epididymitis within the past 3 months.
5. Urethral strictures, bladder neck contracture, unusual anatomy or muscle spasms that would prevent the introduction and use of the Rezūm device.
6. Diagnosed bladder, urethral or ureteral stones or active stone passage in the past 6 months, provided that stones that are known to be in the kidney and have been stable for a period exceeding 3 months are permissible.
7. Subject interested in maintaining fertility.
8. Use of the following medications where the dose is not stable (stable dose defined as the same medication and dose in the last three months):

   1. Beta-blockers;
   2. Anticonvulsants;
   3. Antispasmodics;
   4. Antihistamines;
   5. Alpha blockers for BPH and anticholinergics or cholinergics;
   6. Type II, 5-alpha reductase inhibitor (e.g., finasteride (Proscar, Propecia));
   7. Dual 5-alpha reductase inhibitor (e.g., dutasteride (Avodart));
   8. Estrogen, drug-producing androgen suppression, or anabolic steroids;
   9. PD5 Inhibitors (e.g., Viagra, Levitra or Cialis)
9. Subjects who have had an incidence of spontaneous urinary retention either treated with indwelling transurethral catheter or suprapubic catheter 6 months prior to baseline. A provoked episode now resolved is still admissible
10. Evidence of atonic neurogenic bladder evaluated by a baseline urodynamic assessment.
11. Visible hematuria with subject urine sample without a known contributing factor.
12. Presence of a penile implant or stent(s) in the urethra or prostate
13. Active urinary tract infection by culture within 7 days of treatment or two documented independent urinary tract infections of any type in the past 6 months.

    Gastroenterology:
14. Previous pelvic irradiation or radical pelvic surgery.
15. Previous rectal surgery (other than hemorrhoidectomy) or known history of rectal disease.

    Nephrology:
16. Compromised renal function defined as serum creatinine > 2.0 mg/dl.
17. Hydronephrosis (Grade 2 or higher).

    Oncology:
18. Prostate cancer testing:

    If PSA is > 2.5 ng/ml and ≤ 10 ng/ml with free PSA <25%, prostate cancer for the subject must be/had been ruled out through a negative biopsy prior to enrollment
    * Males 50-59 years - PSA is >2.5 ng/ml and ≤10 ng/ml with free PSA <25%,
    * Males 60+ years - PSA is >4 ng/ml and ≤10 ng/ml, with free PSA <25%
19. History of confirmed malignancy or cancer of the prostate or bladder; however, high grade prostatic intraepithelial "PIN" is acceptable.
20. History of cancer in non-genitourinary system that is not considered cured (except basal cell or squamous cell carcinoma of the skin). A potential participant is considered cured if there has been no evidence of cancer within five years of enrollment.

    Cardiology:
21. History of clinically significant congestive heart failure (i.e., NYHA Class III and IV).
22. Cardiac arrhythmias that are not controlled by medication and/or medical device.
23. An episode of unstable angina pectoris, a myocardial infarction, transient ischemic attack, or a cerebrovascular accident within the past six months.

    Pulmonology:
24. History of significant respiratory disease where hospitalization for the disease is required.

    Hematology:
25. Diagnosed or suspected bleeding disorder, or coagulopathies.
26. Use of antiplatelet or anticoagulant medication except low dose aspirin (<100mg/day) within 10 days prior to treatment.

    Endocrinology:
27. History of diabetes not controlled by a stable dose of medication over the past three months, provided that patients with a hemoglobin A1c <8.0% are allowed.

    Immunology:
28. History of immunosuppressive conditions (e.g., AIDS, post-transplant).

    Neurology:
29. Any cognitive or psychiatric condition that interferes with or precludes direct and accurate communication with the study investigator regarding the study or affect the ability to complete the study quality of life questionnaires.
30. Diagnosed or suspected primary neurologic conditions such as multiple sclerosis or Parkinson's disease or other neurological diseases known to affect bladder function, sphincter function or poor detrusor muscle function (< 25% of accepted and established nomograms).

    General:
31. Currently enrolled in any other pre-approval investigational study in the US (does not apply to long-term post-market studies unless these studies might clinically interfere with the current study endpoints (e.g., limit use of study-required medication, etc.).
32. Any significant medical history that would pose an unreasonable risk or make the subject unsuitable for the study.
33. Inability to provide a legally effective "Informed Consent Form" and/or comply with all the required follow-up requirements.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 47 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Woo, MD, Principal Investigator — Sydney Adventist Hospital
Locations (10):
- United States (9):
  - Arizona Urology Specialists, Scottsdale, Arizona
  - Pinellas Urology, LLC, St. Petersburg, Florida
  - First Urology, PSC, Jeffersonville, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Chesapeake Urology Associates, LLC, Towson, Maryland
  - Adult & Pediatric Urology, P.C., Omaha, Nebraska
  - Jersey Urology Group, Somers Point, New Jersey
  - Houston Metro Urology, Houston, Texas
  - Urology San Antonio, San Antonio, Texas
- Sydney Adventist Hospital/University of Sydney, Wahroonga, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Prostatic Vapor Ablation with Rezum
  Prostatic Vapor Ablation: Rezūm uses the stored thermal energy in water vapor (steam) to treat the extra prostate tissue that is causing symptoms such as frequency, urgency, irregular flow, weak stream, straining and getting up at night to urinate.
  Inside a hand-held device, radiofrequency energy is applied to a few drops of water to create vapor (steam). The water vapor is injected into the prostate tissue that is blocking the flow of urine from the bladder, where it immediately turns back to water, releasing the energy stored in the vapor into the cell membranes. At this point, the cells are gently and immediately damaged, causing cell death. Over time, the body absorbs the treated tissue through its natural healing response.
Period: Overall Study
Arm/Group | Treatment
Started | 47
2 Weeks | 47
6 Weeks | 47
3 Months | 47
6 Months | 47
12 Months | 40
24 Months | 1
Completed | 0
Not Completed | 47
Not completed — Study was terminated for business reasons | 47

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  White | 40
  Hispanic or Latino | 4
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With ≥ 30% Improvement in Symptoms as Measured by the International Prostate Symptom Score (IPSS)
Description: The proportion of the intent-to-treat (ITT) analysis population that responds to the Rezum therapy is reported. A responder is defined as a subject who has an improvement in International Prostate Symptom Score (IPSS) > 30% from baseline to 6 months post-therapy. IPSS scores range from 0 (no symptoms) to 35 (severe symptoms). Improvement in symptoms is shown by a reduction in score.
Time Frame: 6 Months
Population: All subjects enrolled were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 47
Participants | 39

2. Primary Outcome: Number of Participants With Post Procedure Device Related Serious Complications
Description: Assess the composite rate of post procedure device related serious complications in treated subjects through 6 months follow-up.
Time Frame: 6 Months
Population: All subjects enrolled were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 47
Participants | 0

3. Secondary Outcome: Number of Subjects With Device-related Retention Catheterizations
Description: This safety endpoint will be to characterize the rate of post procedure device-related serious retention catheterizations at 6 months.
Time Frame: 6 Month
Population: All subjects enrolled were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 47
Participants | 0

4. Secondary Outcome: Change in Lower Urinary Tract Symptoms as Assessed by the Absolute Change in IPSS Score From Baseline to Follow-up
Description: The change in IPSS from baseline to each follow-up visit was determined. IPSS scores range from 0 (no symptoms) to 35 (severe symptoms). Improvement in symptoms is shown by a reduction in score.
Time Frame: Baseline, 6 weeks, 3 months, 6 months, 1 year
Population: All subjects with data at both baseline and the follow-up visit were included in the analysis (N=47 at 6 weeks, 3 months, 6 months; N=42 at 12 months).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 47
score on a scale
  Change from baseline to 6 weeks post-therapy | -8.47 [-10.49 to -6.45]
  Change from baseline to 3 months post-therapy | -10.97 [-12.68 to -9.27]
  Change from baseline to 6 months post-therapy | -11.62 [-13.43 to -9.80]
  Change from baseline to 12 months post-therapy: number analyzed (Participants) | 42
  Change from baseline to 12 months post-therapy | -11.80 [-13.57 to -10.03]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first patient in until the termination of the study. All 47 subjects were followed to at least the 6- month follow-up visit.
Description: For all adverse events related to the device, the procedure, or the disease state being treated, a Clinical Events Committee was utilized for review and adjudication.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 4/47
Other Adverse Events (participants affected / at risk) | 41/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=47)
Acute Prostatitis (Infections and infestations) | 1 (1) — Acute Prostatitis
Hematuria Gross with Clots & Retention (Renal and urinary disorders) | 1 (1)
Bells Palsy (Nervous system disorders) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) — Worsening of Right Inguinal Hernia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=47)
UTI - Culture Proven (Infections and infestations) | 11 (13)
Hematuria - Gross (Renal and urinary disorders) | 12 (12)
Urinary Urgency (Renal and urinary disorders) | 10 (11)
Bladder Spasms (Renal and urinary disorders) | 10 (10)
Dysuria (Renal and urinary disorders) | 10 (10)
Acute Urinary Retention (Renal and urinary disorders) | 7 (7)
Urinary Incontinence - Urge (Renal and urinary disorders) | 5 (6)
Pain/Discomfort - Other (General disorders) | 4 (5)
Pain/Discomfort - Penile (Reproductive system and breast disorders) | 4 (5)
Poor Stream (Renal and urinary disorders) | 5 (5)
Terminal Dribbling (Renal and urinary disorders) | 4 (4)
Urinary Incontinence - Not Specified (Renal and urinary disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Erectile Dysfunction - Worsening (Reproductive system and breast disorders) | 3 (3)
Nocturia (Renal and urinary disorders) | 3 (3)
Anejaculation (Reproductive system and breast disorders) | 2 (2)
Decrease in Ejaculatory Volume (Reproductive system and breast disorders) | 2 (2)
Epididymitis (Infections and infestations) | 2 (2)
Fever (General disorders) | 2 (2)
Hematospermia (Reproductive system and breast disorders) | 2 (2)
Hesitancy (Renal and urinary disorders) | 2 (2)
Incomplete Voiding (Renal and urinary disorders) | 2 (2)
Sloughing (General disorders) | 2 (2)
Urinary Frequency (Renal and urinary disorders) | 2 (2)
Catheter Malfunction (Product Issues) | 1 (1)
Erectile Dysfunction - De Novo (Reproductive system and breast disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hematuria - Intermittent Uncomplicated (Renal and urinary disorders) | 1 (1)
Hematuria Gross with Clots & Retention (Renal and urinary disorders) | 1 (1)
Pain/Discomfort - Abdominal (Gastrointestinal disorders) | 1 (1)
Pain/Discomfort - Pelvic (Reproductive system and breast disorders) | 1 (1)
Pain/Discomfort - Suprapubic (Reproductive system and breast disorders) | 1 (1)
Retrograde Ejaculation - Confirmed (Reproductive system and breast disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated by the sponsor for business reasons. As a result there is no patient data presented for the 12 month, 2 year and 3 year follow up visits as they did not occur per termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT03605745/Prot_SAP_000.pdf